CLINICAL TRIAL: NCT06158724
Title: COVID-19 Personal Protective Equipment for Vaccinated Health Workers and Convalescents
Status: Withdrawn | Type: Observational
Why Stopped: COVID stopped
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Peter Radsel, asist. prof. Peter Radšel, MD, PhD., Head of intensive internal medicine department, University Medical Centre Ljubljana
Other Study IDs: CIIM-KIBVS COVID
Record Dates: First submitted 2023-12-05; First posted 2023-12-06 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Covid19
Keywords: Covid19; SARS-CoV 2; Personal Protective Equipment; Safety
MeSH Terms: conditions — COVID-19 | interventions — Personal Protective Equipment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Simplified PPE group: Surgical mask, standard non sealing goggles, use of protective gown while in direct contact with patients.
  Interventions: Other: Personal Protective Equipment
- Standard COVID-19 PPE: FFP2 mask, goggles and face shield, protective gown for COVID-19 ward.
  FFP 3 mask or filter gas mask, sealing goggles, face shield or hazmat suit, protective gown, gloves and surgical cap.

INTERVENTIONS:
Other: Personal Protective Equipment — Simplified PPE for use in COVID-19 departments.
  Groups: Simplified PPE group

SUMMARY:
The aim of the trial is to assess the safety of using simplified personal protective equipment (PPE) for vaccinated or COVID-19 convalescent healthcare workers working in COVID-19 ICU or COVID-19 wards.

The trial is designed as a prospective randomized observational trial with volunteer medical staff working in COVID-19 departments aiming to show non-inferiority of simplified PPE vs standard COVID-19 PPE.

DETAILED DESCRIPTION:
Objectives To assess safety of simplified personal protective equipment (PPE) for vaccinated health workers and COVID-19 convalescents - pilot trial.

Methods Prospective randomized observational trial. 60 participants randomized 1:1 to either standard PPE (COVID-19 ward: FFP2 or higher respirator, goggles of face shield, gown, gloves; COVID-19 ICU: FFP3 respirator and tight goggles or full face mask or powered air-purifying respirators, gown and gloves) or simplified PPE (surgical mask, goggles or face shield, gown). 30 days follow up period.

Participants Volunteer medical staff from COVID-19 regular and ICU departments at University Medical Center Ljubljana, Slovenia, with either proven COVID-19 infection within 6 months or at least 7 days after second dose anti COIVD-19 vaccine.

Hypotheses Simplified PPE is non-inferior to standard PPE in vaccinated health workers or convalescents.

Discussion Positive study results may decrease PPE spending cost and positively affect working conditions at COVID-19 departments.

ELIGIBILITY:
Inclusion Criteria:

* age < 50 years
* prior COVID-19 infection; time from infection < 6 months.
* prior completed anti COVID-19 immunization; > 1 week post second dose of immunization.
* signed written consent
* negative nasopharyngeal COVID-19 RT-PCR test

Exclusion Criteria:

* age > 50 years
* time post COVID-19 infection > 6 months
* time post COVID-19 immunization < 1 week.
* immunocompromised patients
* pregnancy
* CKD 3 or more
* COPD or other lung disease
* heart failure of any cause
* ischemic heart disease
* obesity (BMI > 30)
* DM on therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteer healthy healthcare workers working in COVID-19 departments.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of simplified PPE compared to standard PPE regarding symptomatic infection rate. | 30 days
  The use of simplified PPE will not predispose COVID-19 immune healthcare workers to symptomatic neoinfection.

SECONDARY OUTCOMES:
Non-inferiority of simplified PPE compared to standard PPE regarding asymptomatic infection rate. | 30 days
  No difference in nasopharyngeal RT-PCR SARS-CoV 2 results between groups.
Rise in anti-SARS-CoV 2 antibody titers in the simplified PPE group. | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gross JV, Mohren J, Erren TC. COVID-19 and healthcare workers: a rapid systematic review into risks and preventive measures. BMJ Open. 2021 Jan 20;11(1):e042270. doi: 10.1136/bmjopen-2020-042270. PMID 33472783
- [Background] Sewell HF, Agius RM, Kendrick D, Stewart M. Covid-19 vaccines: delivering protective immunity. BMJ. 2020 Dec 17;371:m4838. doi: 10.1136/bmj.m4838. No abstract available. PMID 33334862
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Widge AT, Rouphael NG, Jackson LA, Anderson EJ, Roberts PC, Makhene M, Chappell JD, Denison MR, Stevens LJ, Pruijssers AJ, McDermott AB, Flach B, Lin BC, Doria-Rose NA, O'Dell S, Schmidt SD, Neuzil KM, Bennett H, Leav B, Makowski M, Albert J, Cross K, Edara VV, Floyd K, Suthar MS, Buchanan W, Luke CJ, Ledgerwood JE, Mascola JR, Graham BS, Beigel JH; mRNA-1273 Study Group. Durability of Responses after SARS-CoV-2 mRNA-1273 Vaccination. N Engl J Med. 2021 Jan 7;384(1):80-82. doi: 10.1056/NEJMc2032195. Epub 2020 Dec 3. No abstract available. PMID 33270381